CLINICAL TRIAL: NCT05915052
Title: A New Type of Temporary Ileostomy --B-suture Ileostomy Applied to Laparoscopic Low Anterior Rectal Resection
Brief Title: B-suture Ileostomy in Clinical Practice: a Retrospective, Single-center, Propensity Score-matched Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Daorong Wang, DR, Northern Jiangsu People's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NorthernJiangsu002
Record Dates: First submitted 2023-06-05; First posted 2023-06-22 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Ileostomy; Ileostomies; Loop Ileostomies
Keywords: Loop Ileostomies; ileostomy; traditional; laparoscopic low anterior rectal resection; complications

STUDY DESIGN:
Intervention Model Description: To minimize bias in baseline characteristics between the B-suture stoma group and the conventional method stoma group, we performed propensity score matching (pSM) with a matching tolerance (M) set at 0.02 and nearest neighbor matching without put-back at a ratio of 1:1. Baseline information for matching was: gender, age, BMI, hemoglobin, albumin, diabetes, hypertension, previous abdominal surgery history, distance of the lower margin of the tumor from the anal margin, tumor diameter, American Society of Anesthesiology (ASA) physical classification, and tumor stage. 62 patients in the B-suture stoma group were successfully matched 1:1 with 123 patients in the conventional stoma group to 59 patients in the B-suture stoma group and 59 patients in the conventional stoma group. 59 patients in the B-stitch stoma group and 59 patients in the conventional stoma group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the B-type suture ileostomy group (Active Comparator): the B-type suture ileostomy group underwent laparoscopic low anterior resection and a B-type suture ileostomy
  Interventions: Procedure: B-type suture ileostomy
- the traditional ileostomy group (Active Comparator): the traditional ileostomy group underwent laparoscopic low anterior resection and a traditional ileostomy
  Interventions: Procedure: the traditional ileostomy

INTERVENTIONS:
Procedure: B-type suture ileostomy — Type B suture stoma group：2-0 stitched sutures were placed in the center of the incision, from the anterior rectus sheath on the left side of the incision → the posterior rectus sheath on the left side of the incision → through the avascular area below the vascular arch at the mesenteric border of the ileum to the contralateral side → the posterior rectus sheath on the right side of the incision → the anterior rectus sheath on the right side of the incision→ the posterior rectus sheath on the right side of the incision → through the avascular area below the vascular arch at the mesenteric border of the ileum to the contralateral side → the posterior rectus sheath on the left side of the incision →the anterior rectus sheath on the left side of the incision sutures were sewn through in the sequence, tightened and knotted .
  Arms: the B-type suture ileostomy group
Procedure: the traditional ileostomy — Then take the right lower abdominal incision to cut a circular incision of 3 cm in diameter, round excision of subcutaneous fat, cross incision of rectus sheath and peritoneum, enter the abdomen, raise the marked ileum out of the body, interrupt suture of ileum with peritoneum and posterior sheath of rectus abdominis for one week, then interrupt suture of ileum with anterior sheath of rectus abdominis for one week, transverse incision of 2 cm in diameter, interrupted with 3-0 absorbable thread, The ileocecal incision and the skin of the right lower abdominal circular incision were sutured for one week to complete the double-lumen stoma at the end of the ileum.
  Arms: the traditional ileostomy group

SUMMARY:
OBJECTIVE: The purpose of this study was to introduce a new temporary ileostomy modality, the B-suture ileostomy, and to compare its technical advantages in comparison with conventional ileostomy.

CONCLUSION: This study shows that B-suture ileostomy can simplify the surgical procedure, facilitate learning and promotion, shorten the stoma and surgical time, can reduce complications such as irritant dermatitis, peristoma infection, stoma stricture, stoma retraction, shorten the hospital stay, reduce postoperative pain, and is similar to the traditional procedure in terms of secondary surgical return, which is a surgical procedure worth continuing to explore.

DETAILED DESCRIPTION:
OBJECTIVE: The purpose of this study was to introduce a new temporary ileostomy modality, the B-suture ileostomy, and to compare its technical advantages in comparison with conventional ileostomy.

METHODS: A retrospective single-center study analyzed 185 patients undergoing laparoscopic low anterior resection for rectal cancer combined with temporary ileostomy, collecting general case data, surgery-related data, postoperative-related complications, secondary surgical return data, and postoperative health status data, and divided into a B-suture ileostomy group (n=62) and a conventional method ileostomy group (n=123) according to the different stoma methods, by propensity score matching (pSM) for 1:1 matching (n=59 for both groups after matching). The advantages and disadvantages of the B-suture method ileostomy were evaluated by analyzing and comparing information on the perioperative period, postoperative related complications, and postoperative health status.

ELIGIBILITY:
Inclusion Criteria:

* If necessary, combine bulleted, numbered, and lettered lists in order to create lists within a list. For example:simultaneous laparoscopic low anterior resection of rectal cancer + temporary ileostomy;
* pathologically confirmed primary rectal cancer;
* rectal tumor height ≤12 cm from the anal verge;
* no tumor metastasis at the time of surgical resection;
* all surgeries were performed by the same surgical team with more than 10 years of experience in laparoscopic radical resection of rectal cancer and ileostomy.

Exclusion Criteria:

* patients who did not undergo stoma rejection due to tumor metastasis or recurrence;
* patients who were too old or in poor general condition to undergo stoma reversal surgery;
* patients with multiple primary colorectal cancers who underwent simultaneous multifocal resection;
* patients with incomplete clinical medical information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
total operative time | one year
  the operating time of the two groups
ileostomy time | one year
  time spent on ileostomies by the two groups
bleeding volume | one year
  Intraoperative bleeding in both groups
time of stoma evacuation | one year
  time of stoma evacuation for the two groups
time of starting to eat | one year
  time of starting to eat in both groups
time to first ambulation | one year
  time to first ambulation in both groups
postoperative hospital stay | one year
  postoperative hospital stay in both groups

SECONDARY OUTCOMES:
Complications related to the stoma | one year
  Complications related to the stoma in both groups，such as irritant dermatitis、Parastomal hernia、Incisional hernia、Intestinal obstruction、Stoma bleeding Peristomal infection、Infection of specimen 、removal incision、Stoma stenosis、Stoma retraction、Stoma prolapse、Dehydration

CONTACTS AND LOCATIONS:
Overall Officials: sun longhe, Master, Principal Investigator — https://www.yzsbh.com/
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun L, Zhou J, Ji L, Wang W, Zhang Q, Qian C, Zhao S, Li R, Wang D. Clinical application of the B-type sutured ileostomy in robotic-assisted low anterior resection for rectal cancer: a propensity score matching analysis. J Robot Surg. 2024 Apr 5;18(1):159. doi: 10.1007/s11701-024-01924-8. PMID 38578352